CLINICAL TRIAL: NCT02135055
Title: Effect of Midazolam on Inflammatory Response and Organ Function in Mechanically Ventilated Sepsis Patients With Different Immune Status.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014021801
Record Dates: First submitted 2014-04-29; First posted 2014-05-09 (Estimated); Last update posted 2014-05-09 (Estimated); Status verified 2014-05

CONDITIONS: Inflammatory Disorder of Immune System; Sepsis
Keywords: organ function; sedation
MeSH Terms: conditions — Sepsis | interventions — Midazolam; Morphine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Normal immune function (Experimental): The value of monocyte human leukocyte antigen-DR (mHLA-DR) is equal to or more than 15000 monoclonal antibody.
  Interventions: Other: blood sample collection; Drug: Midazolam; Drug: Morphine; Procedure: Sedation interruption
- Moderate immunosuppression (Experimental): The value of mHLA-DR is equal to or more than 10000 and less than 15000 monoclonal antibody.
  Interventions: Other: blood sample collection; Drug: Midazolam; Drug: Morphine; Procedure: Sedation interruption
- Sever immunosuppression (Experimental): The value of mHLA-DR is equal to or more than 5000 and less than 10000 monoclonal antibody.
  Interventions: Other: blood sample collection; Drug: Midazolam; Drug: Morphine; Procedure: Sedation interruption
- Immune paralysis (Experimental): The value of mHLA-DR is less than 5000 monoclonal antibody.
  Interventions: Other: blood sample collection; Drug: Midazolam; Drug: Morphine; Procedure: Sedation interruption

INTERVENTIONS:
Other: blood sample collection — Patients were included 1 hrs later(before the study drug is administrated), 3 d and 7 d after sedation with midazolam, blood sample is collected. Flow cytometry is performed to test the mHLA-DR and according the value of mHLA-DR, assign the participant to the 4 groups as described in the arm.
Drug: Midazolam — The loading dose of midazolam is 0.03-0.3 mg/kg, intravenous injected slowly for 10 minutes, then 0.04-0.2 mg/kg/h for maintenance of sedation.
  Other Names: Liyuexi
Drug: Morphine — Morphine is the only analgesic drug that permitted to use. 2 mg morphine is given a bolus when the participant feel pain. If the pain is not alleviated, 0.4-1 mg/h morphine is maintained.
Procedure: Sedation interruption — Sedation interruption is performed at 8 am every morning.

SUMMARY:
ICU patients always experience all kinds of pain, discomfort and sleep disturbance,especially the sepsis patients. Appropriate sedation and analgesia is must,the newest sepsis guideline strongly recommend that mechanically ventilated sepsis patients need sedation therapy.

Recent studies show than immune dysfunction dose have an important effect on the occurrence and development of sepsis. When the body suffer from the pathogenic microorganism attacking and sepsis, it activate the systemic inflammatory response (SIRS) and compensatory anti-inflammatory response syndrome (CARS). When it is out of balance between SIRS and CARS, the inflammatory response, immune paralysis or immune dysfunction occurs and the mixed anti-inflammatory response syndrome (MARS) exists, and then the multiple organ dysfunction. So, immune dysfunction is thought to be the key factors on the development of the sepsis. Some studies show that the sedation drug such as midazolam, propofol, dexmedetomidine could suppress the inflammatory response effectively and then modulate the immune function.

Several recent studies show that midazolam has the immunoregulation effect and trend of suppress the inflammatory response, but the result is controversy, the possibly reason is the different immune status. Now there is the guideline about the different immune status: the normal immune function means that the value of mHLA-DR is more than 15000 monoclonal antibody; moderate-sever immune suppression means that the value of mHLA-DR is in the range of 5000 and 15000 monoclonal antibody; the immune paralysis means that the value of mHLA-DR is less than 5000 monoclonal antibody.

The purpose of the study is to explore the effect of midazolam to inflammatory response and organ function at mechanically ventilated sepsis patients who have different immune status.

ELIGIBILITY:
Inclusion Criteria:

1. Mechanically ventilated ICU patients, sedation is needed.
2. Sepsis patients.
3. Age 18-80 yrs
4. Anticipated sedation duration is more than 3 days.
5. Agreed to participate the study and assigned the informed consent. -

Exclusion Criteria:

1. Allergic to the Benzodiazepine.
2. Hepatic dysfunction(Child-Pugh is C level).
3. Participated other study.
4. Bad prognosis and possibly become the major reason of patients death, such as sever craniocerebral injury,cardiopulmonary resuscitation,advanced malignant tumor,etc.
5. History of immune system disease, immune treatment (including hormone ) or treatment that could affect immune function (including continuous renal replacement therapy,CRRT).
6. Alcoholic and drug abuse.
7. Tendency for major mental disease or treatment of anti psychotics.
8. Pregnant,lactation woman.
9. Unwilling to assign the informed consent or bad compliance. -

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2014-05; Primary Completion 2015-03 (Estimated); Study Completion 2015-03 (Estimated)

PRIMARY OUTCOMES:
T cell subset T Helper 1 | Change from baseline of T Helper 1 at 3 and 7 days.
  T Helper 1(TH1) are tested before sedation, 3 d and 7 d after sedation with midazolam.
  The test method is Flow cytometry.
T cell subset T Helper 2 | Change from baseline of T Helper 2 at 3 and 7 days.
  T Helper 2(TH2) are tested before sedation, 3 d and 7 d after sedation with midazolam.
  The test method is Flow cytometry.
T cell subset Regulatory T Cell | Change from baseline of Regulatory T Cell at 3 and 7 days.
  Regulatory T Cell are tested before sedation, 3 d and 7 d after sedation with midazolam.
  The test method is Flow cytometry.
Interleukin-6 | Change from baseline of Interleukin-6 at 3 and 7 days.
  Levels of interleukin-6(IL-6) are tested before sedation, 3 d and 7 d after sedation with midazolam.
  The test method is Enzyme Linked Immunosorbent Assay（ELISA）.
Interleukin-10 | Change from baseline of Interleukin-10 at 3 and 7 days.
  Levels of interleukin-10(IL-10) are tested before sedation, 3 d and 7 d after sedation with midazolam.
  The test method is Enzyme Linked Immunosorbent Assay（ELISA）.
Tumo necrosis factor-α(TNF-α) | Change from baseline of TNF-α at 3 and 7 days.
  Levels of Tumo necrosis factor-α(TNF-α) are tested before sedation, 3 d and 7 d after sedation with midazolam.
  The test method is Enzyme Linked Immunosorbent Assay（ELISA）.

SECONDARY OUTCOMES:
duration of mechanical ventilation | from the begining of ventilation to weaning, up to 7 days.
Number of Participants with Serious and Non-Serious Adverse Events | up to 7 days
Mortality | up to 28 days
  Participants' mortality of 28 and 90 days is recorded, including state of survival, the date and the reason of death.
Length of ICU stay | from ICU admmittion to discharge from ICU,up to 28 days.
Index of renal function | baseline,the 3rd and 7th day after sedation
  level of Blood Urea Nitrogen(BUN) and Creatinine(Cr).
Index of myocardial enzyme | baseline,the 3rd and 7th day after sedation
  level of Brain Natriuretic Peptide(BNP).
Index of hepatic function | baseline,the 3rd and 7th day after sedation
  level of glutamic-pyruvic transaminase(ALT),glutamic oxalacetic transaminase(AST),Total Bilirubin(Tbil).
Index of endocrine function | baseline,the 3rd and 7th day after sedation
  level of cortisol and blood glucose.
C-reaction protein | baseline,the 3rd and 7th day after sedation
  C-reaction protein(CRP)is tested before sedation, 3 d and 7 d after sedation with midazolam.
  The test method is Enzyme Linked Immunosorbent Assay（ELISA）.

OTHER OUTCOMES:
mHLA-DR | baseline,the 3rd and 7th day after sedation
  Levels of mHLA-DR are tested before sedation, 3 d and 7 d after sedation with midazolam.
  The test method is Flow cytometry.

CONTACTS AND LOCATIONS:
Overall Officials: Yuhang Ai, Doctor., Principal Investigator — Xiangya Hospital of Central South University